CLINICAL TRIAL: NCT00746239
Title: Ramelteon for Sleep Initiation Insomnia in Panic Disorder Who Are Also on Escitalopram for Anxiety: A Double Blind, Randomized Clinical Trial
Brief Title: Ramelteon for Sleep Initiation Insomnia in Individuals With Panic Disorder Who Are Also on Escitalopram for Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for continuation was not received.
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-013R
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Panic Disorder; Insomnia
Keywords: insomnia; sleep difficulty; panic disorder; nocturnal panic attacks; anxiety
MeSH Terms: conditions — Panic Disorder; Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Escitalopram; ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Subjects will be randomly assigned to receive either Ramelteon and Escitalopram OR Placebo and Escitalopram.
  Interventions: Drug: Ramelteon and Escitalopram
- 2 (Placebo Comparator): Subjects will be randomly assigned to receive either Ramelteon and Escitalopram OR Placebo and Escitalopram.
  Interventions: Drug: Placebo and Escitalopram

INTERVENTIONS:
Drug: Placebo and Escitalopram — Placebo and Escitalopram (5 to 40 mg)
  Arms: 2
Drug: Ramelteon and Escitalopram — Ramelteon 8 mg and Escitalopram (5-40 mg)
  Arms: 1

SUMMARY:
Almost 80% of panic disorder patients report difficulty sleeping. Sleep disturbances in turn may exacerbate underlying anxiety/panic attacks. Moreover, individuals with insomnia (sleep disturbance) are at higher risk of developing a new anxiety disorder. Therefore it is expected that improving sleep quality with medications along with other medications to treat anxiety component of panic disorder might be helpful. However, there is lack of pharmacological studies examining the effects of improving sleep disturbances with medications in panic disorder patients, which is a critical problem for providing optimal care to these patients. The objective of this proposal is to determine the effects of ramelteon (FDA approved for insomnia) on sleep disturbances in Panic disorder patients who are on escitalopram for underlying anxiety.

ELIGIBILITY:
Inclusion Criteria:

* 1) Clinical diagnosis of panic disorder
* 2) Difficulty initiating sleep (subjective sleep latency (SL) of >30 minutes) for at least 3 times per week in the preceding month.

Exclusion Criteria:

* 1)Patients meeting DSM-IV criteria (as determined by MINI) for a current anxiety disorder (other than panic disorder), or current major depressive disorder that is considered by the investigator to be primary (i.e., causing a higher degree of distress or impairment than panic disorder)., Patients with past history of DSM-IV anxiety disorders or depressive disorder will not be excluded.
* 2) Patients with current psychotic disorder, current bipolar disorder, or substance use disorder (except nicotine dependence) or Subjects with significant suicide risk.
* 3) Candidates with known sensitivity to any selective serotonin reuptake inhibitors (SSRI) will be excluded.
* 4) CNS diseases: Candidates with seizure disorder (other than febrile seizure in early childhood), a history of other neurological disorder, and head trauma will be excluded.
* 5) Cardiovascular and respiratory diseases: Candidates with hypertension (systolic >130; diastolic > 85), arrhythmias, coronary artery disease, cardiac pacemakers, COPD, asthma, and other pulmonary diseases will be excluded.
* 6) Primary sleep disorders: Candidates with breathing related sleep disorder, restless leg syndrome, circadian rhythm sleep disorders, narcolepsy, and other major primary sleep disorders will be excluded.
* 7) Systemic diseases: Candidates with other medical problems, such as endocrinopathies, renal or hepatic failure, autoimmune diseases involving the CNS, obesity (BMI > 30 kg/m2), or a history of pheochromocytoma will not be eligible.
* 8) Consumption of greater than 720 mgs. of caffeine daily.
* 9) History of shift work (11 PM to 7 AM) in the past 6 months.
* 10) Reproductive status: Women candidates who are pregnant (based on urine test) are not eligible. Women of child bearing age will be on birth control methods during the study period.
* 11) Individuals with personality, behavior, or medical disorders likely to interfere with study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Singareddy, MD, Principal Investigator — Penn State College of Medicine/Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- See also: National Institute of Mental Health Patient information page — http://www.nimh.nih.gov/health/topics/panic-disorder/index.shtml
- See also: American Medical Association Medem links to panic disorder — http://www.medem.com/MedLB/article_detaillb.cfm?article_ID=ZZZXHSH3DMC&sub_cat=47
- See also: MedlinePlus panic disorder information — http://www.nlm.nih.gov/medlineplus/panicdisorder.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects total were enrolled in the study. It was a double blind study, however, the blind was never opened as the study was terminated prematurely due to lack of continued funding. Thus, subjects in each arm are not known. Out of the 11 subjects enrolled, 6 withdrew from the study and 5 completed the study.
Groups:
- PD Subjects With Either Escitalopram and Placebo OR Ramelteon: Subjects were randomly assigned to receive either Ramelteon 8 mg and Escitalopram (5-40 mg) OR Placebo and Escitalopram (5-40 mg). However, as the blind was never opened, we are combining all subjects in one group for presenting in this record.
Period: Overall Study
Arm/Group | PD Subjects With Either Escitalopram and Placebo OR Ramelteon
Started | 11
Completed | 5 (11 subjects total were enrolled - 6 withdrew from study and 5 competed)
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- PD Subjects With Either Escitalopram and Placebo OR Ramelteon: Panic disorder subjects who were on Escitalopram (5-40 mg) received either Ramelteon 8 mg OR Placebo. As the study was terminated prematurely, the blind was never opened. Thus, it is not known as to how many were in each arm. As a result we are combining all subjects in one group for presenting in this record.
Arm/Group | PD Subjects With Either Escitalopram and Placebo OR Ramelteon
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effects of Ramelteon on Sleep Quality in Panic Disorder Patients Who Are Also Treated With Escitalopram.
Time Frame: 10 weeks
Groups:
- PD Subjects With Either Escitalopram and Placebo OR Ramelteon: 11 subjects enrolled- 6 withdrew from study/the blind was never opened as the study was terminated prematurely for lack of continued funding- the data for outcome measures was never collected/compiled/analyzed
Arm/Group | PD Subjects With Either Escitalopram and Placebo OR Ramelteon
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Association of Improving Sleep Quality (With Ramelteon) on Improvement in Severity of Panic Disorder/Anxiety.
Time Frame: 10 weeks
Arm/Group | PD Subjects With Either Escitalopram and Placebo OR Ramelteon
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years 2 months
Groups:
- PD Subjects With Either Escitalopram and Placebo OR Ramelteon: Panic disorder subjects who were on Escitalopram received either Escitalopram OR Placebo - as the study terminated prematurely, the blind was never opened; thus it is not known as to how many were in each arm- as a result we are not combining all in one group for presenting in this record.
  Ramelteon and Escitalopram: Ramelteon 8 mg and Escitalopram (5-40 mg)
Arm/Group | PD Subjects With Either Escitalopram and Placebo OR Ramelteon
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PD Subjects With Either Escitalopram and Placebo OR Ramelteon (N=11)
extreme drowsiness and difficult focussing (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes